CLINICAL TRIAL: NCT03232164
Title: PSMA-based 18F-DCFPyL PET/CT and PET/MRI Pilot Studies in Prostate Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UW16062; 2016-0883 (Other: Institutional Review Board); A539300 (Other: UW Madison); NCI-2017-01643 (Registry Identifier: NCI Trial ID); Protocol Version 8/25/2023 (Other: UW Madison); Bluemke Family Trust (Other: Private)
Record Dates: First submitted 2017-07-17; First posted 2017-07-27 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer; Prostate Neoplasm
Keywords: Prostate Cancer; Prostate neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single center, open label, single-arm, pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-DCFPyL PET (Experimental): Four separate substudies evaluating 18F-DCFPyL PET imaging of prostate cancer in four prostate cancer clinical scenarios under the following subheadings: (1) primary prostate cancer, (2) biochemical recurrence post-prostatectomy prior to radiation therapy, (3) androgen-resistant metastatic disease and (4) detection of clinically significant prostate cancer in low to intermediate risk primary prostate cancer
  Interventions: Drug: 18F-DCFPyL PET

INTERVENTIONS:
Drug: 18F-DCFPyL PET — 18F-DCFPyL PET demonstrates very high tumor-to-background and tumor specific uptake which may allow for a more sensitive and accurate method for detection of early tumor recurrence and metastatic disease as compared to current PET radiotracers and current standard-of-care imaging including 99mTc-methylene diphosphonate bone scintigraphy (bone scan), contrast-enhanced computed tomography (CT) and magnetic resonance imaging (MRI).

SUMMARY:
The overall goal of this research is to validate and develop a non-invasive imaging biomarker of prostate cancer detection, progression, and recurrence. Development of such a biomarker may be useful to differentiate indolent from aggressive prostate cancer phenotypes allowing for selection of an appropriate risk adaptive therapy.

DETAILED DESCRIPTION:
The investigators propose to evaluate a novel second-generation low-molecular-weight prostate specific membrane antigen (PSMA)-based positron emission tomography (PET) agent, 18F-DCFPyL, for detection of primary and metastatic prostate cancer. 18F-DCFPyL PET demonstrates very high tumor-to-background and tumor specific uptake which may allow for a more sensitive and accurate method for detection of early tumor recurrence and metastatic disease as compared to current PET radiotracers and current standard-of-care imaging including 99mTc-methylene diphosphonate bone scintigraphy (bone scan), contrast-enhanced computed tomography (CT) and magnetic resonance imaging (MRI).

Primary Objectives: The investigators propose to evaluate this PET agent for four different prostate cancer clinical scenarios.

1. detection of clinically significant high-grade prostate cancer and initial staging
2. detection of sites of recurrence in the setting of biochemical recurrence after definitive prostatectomy
3. detection of advanced androgen-resistant metastatic prostate cancer, and
4. detection of clinically significant prostate cancer in very low to intermediate risk primary prostate cancer

Secondary Objectives:

* Evaluate the performance of 18F-DCFPyL PET and MRI whole body DWI for detection of local-nodal and distant metastatic disease on initial staging compared to conventional imaging modalities (CT and bone scintigraphy).
* Correlate 18F-DCFPyL PET standardized-uptake values (SUV) and MRI parameters with PSMA expression by prostatectomy pathology IHC.
* Evaluate the specificity of 18F-DCFPyL PET for differentiating primary prostate cancer versus non-malignant prostate lesions (BPH, prostatitis).
* Comparison of whole body low-dose CT and whole body MRI derived PET SUV-quantitation.
* Evaluate the performance of dedicated pelvic 18F-DCFPyL PET/MRI with dynamic PET acquisition and multi-parametric MRI for differentiation of urine versus recurrent malignancy in the prostatectomy bed.
* Evaluate the contribution of whole body MRI DWI obtained from PET/MRI to improve the diagnostic performance of 18F-DCFPyL PET/CT and PET/MRI for metastatic prostate cancer lesion detection.
* Assess the quantitative accuracy of PET-derived standardized uptake value (SUV)-based parameters in 18F-DCFPyL PET obtained from PET/MRI versus PET/CT.
* Assess the quantitative reproducibility of 18F-DCFPyL PET/CT derived-SUV values in normal organ and metastatic tumor lesions.
* Evaluate the ability of 18F-DCFPyL PET to improve detection of clinically significant primary prostate cancer in men with very low to intermediate risk prostate cancer under active surveillance or watchful waiting.

Update: As of July 2022 verification, the investigators are no longer enrolling into sub-studies 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer pathologically proven by prostate biopsy (newly diagnosed for Sub-Study 1 and 4)
* Prostate biopsy histology grade ≥ Gleason 1, 6, 3+4, or 4+3; positive biopsy >2 cores
* Any PSA permitted
* Two consecutive rising PSA values (Sub-Study 3 only)
* Castrate-levels of testosterone - total testosterone < 50 ng/dL (Sub-Study 3 only)
* Patients considered as candidates for and medically fit to undergo prostatectomy
* At least 7 days after most recent prostate biopsy
* Imaging evidence of suspected metastatic disease, including CT, bone scan, MRI, ultrasound or other PET modalities (Sub-Study 3 only)
* New diagnosis of prostate cancer undergoing additional biopsy evaluation (Sub--Study 4 only)
* Karnofsky performance status of at least 70 (Sub-Study 4 only)
* General health and anatomy suitable to undergo transrectal ultrasound-MRI fusion biopsy of the identified lesions and standard 12 core sextent biopsy (Sub-Study 4 only)

Exclusion Criteria:

* Prior pelvic external beam radiation therapy or brachytherapy
* Chemotherapy for prostate cancer
* Androgen deprivation therapy for prostate cancer
* Investigational therapy for prostate cancer (Sub-Study 3 Only)
* Unable to lie flat during or tolerate PET/CT
* Prior history of any other malignancy within the last 2 years, other than skin basal cell or cutaneous superficial squamous cell carcinoma that has not metastasized and superficial bladder cancer.
* No prostatectomy scheduled more than 12 hours post imaging (Sub-Study 1 only)
* Serum creatinine > 2 time the upper limit of normal
* Total bilirubin > 3 times the upper limit of normal
* Liver Transaminases > 5 times the upper limit of normal

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
18F-DCFPyL PSMA-based PET and multi-parametric MRI with DWI for Sub-Study 1: Primary Prostate Cancer | one study visit (up to 3.5 hours)
  To evaluate the performance of 18F-DCFPyL PSMA-based PET and multi-parametric MRI (MP-MRI) with DWI (Diffusion Weighted Imaging) and gadolinium DCE (Dynamic Contrast Enhanced) using a dedicated PET/MRI scanner to detect clinically significant larger volume high-grade primary prostate cancer based on prostatectomy step-section pathology correlation.
Evaluate 18F-DCFPyL PSMA-based PET for localization for Sub-Study 2: Biochemical Recurrence | one study visit (up to 3.5 hours)
  To evaluate the performance of 18F-DCFPyL PSMA-based PET for localization of the site of recurrent prostate cancer in men with biochemical recurrence after definitive prostatectomy with planned salvage external-beam radiation therapy (EBRT). PSA response to prostatic fossa salvage irradiation will be compared with pre-salvage 18F-DCFPyL PET uptake in the radiation field.
Compare detectability of 18F-DCFPyL for Sub-Study 3: Metastatic Androgen-Resistant Prostate Cancer | up to 7 days
  To compare the detectability of metastatic prostate cancer using 18F-DCFPyL PET obtained from PET/CT and PET/MRI compared to conventional imaging modalities (CIM) (bone scan and CT) in men with androgen-resistant prostate cancer.
Sub-Study 4: Rate of positive cancer detection using PET/MRI directed MRI/transrectal ultrasound (TRUS) fusion biopsy with and without additional PSMA PET information | one study visit (up to 3.5 hours)
  To evaluate the ability of 18F-DCFPyL PSMA PET to improve detection of clinically significant cancer in men with very low to intermediate risk prostate cancer using a dedicated PET/MRI.

SECONDARY OUTCOMES:
Sub-study 1: Detection of local-nodal and distant metastatic disease (PET | one study visit (up to 3.5 hours)
  Evaluate the performance of 18F-DCFPyL PET and MRI whole body DWI for detection of local-nodal and distant metastatic disease on initial staging compared to conventional imaging modalities (CT and bone scintigraphy).
Sub-Study 1: Correlation of 18F-DCFPyL PET and MRI | one study visit (up to 3.5 hours)
  Correlate 18F-DCFPyL PET standardized-uptake values (SUV) and MRI parameters with PSMA expression by prostatectomy pathology IHC.
Sub-Study 1: Specificity of 18F-DCFPyL | one study visit (up to 3.5 hours)
  Evaluate the specificity of 18F-DCFPyL PET for differentiating primary prostate cancer versus non-malignant prostate lesions (BPH, prostatitis).
Sub-Study 1: Low-dose CT versus MRI derived PET SUV | one study visit (up to 3.5 hours)
  Comparison of whole body low-dose CT and whole body MRI derived PET SUV-quantitation.
Sub-Study 2: Detection of local-nodal and distant metastatic disease (pelvic) | one study visit (up to 3.5 hours)
  Comparison of whole body 18F-DCFPyL PET with pelvic MR-MRI and whole body DWI for detection of local-nodal and distant metastatic disease on initial staging compared to conventional imaging modalities (CT and bone scintigraphy).
Sub-Study 2: Dedicated pelvic 18F-DCFPyL PET/MRI with dynamic PET acquisition and multi-parametric MRI | one study visit (up to 3.5 hours)
  Evaluate the performance of dedicated pelvic 18F-DCFPyL PET/MRI with dynamic PET acquisition and multi-parametric MRI for differentiation of urine versus recurrent malignancy in the prostatectomy bed.
Sub-Study 3: Contribution of whole body MRI DWI | Up to 7 days
  Evaluate the contribution of whole body MRI DWI obtained from PET/MRI to improve the diagnostic performance of 18F-DCFPyL PET/CT and PET/MRI for metastatic prostate cancer lesion detection.
Sub-Study 3: Quantitative accuracy | Up to 7 days
  Assess the quantitative accuracy of 18F-DCFPyL PET standardized uptake value parameters from PET/MRI versus PET/CT.
Sub-Study 3: Quantitative reproducibility | Up to 7 days
  Assess the quantitative reproducibility of 18F-DCFPyL PET/CT derived-SUV values in normal organ and metastatic tumor lesions.
Sub-study 4: Positive Detection Rate of Prostate Cancer via biopsy on PSMA PET versus mpMRI alone in very low to intermediate risk groups active surveillance and watchful waiting patients | one study visit (up to 3.5 hours)
  Evaluate the positive detection rate of prostate cancer via biopsy on PSMA PET versus mpMRI alone in very low to intermediate risk groups active surveillance and watchful waiting patients.
Sub-study 4: Detection rate of clinically significant prostate cancer in men with directed MRI/US biopsy | one study visit (up to 3.5 hours)
  To evaluate the ability of PSMA PET alone versus mpMRI alone versus combined PSMA PET with mpMRI to detect clinically significant prostate cancer in men with directed MRI/US biopsy.
Sub-study 4: Detection Rate of Prostate Cancer vs False Positive Findings via Biopsy | one study visit (up to 3.5 hours)
  Evaluate the rate of detection of prostate cancer and false positive findings via biopsy and available prostatectomy histopathology on PSMA PET/MRI versus mpMRI alone in different prostate anatomic regions (transition, central, peripheral zones) in these risk cohorts.
Sub-study 4: Number of Participants who change treatment and surgical management plans after inclusion of PSMA-based PET directed biopsy | one study visit (up to 3.5 hours)
  Assess the change in treatment and surgical management plan before and after inclusion of PSMA-based PET directed biopsy histopathology information and additional pelvic and whole body PET/MRI PET information will be obtained.
Sub-study 4: Correlation of PET and MRI parameters for PET and/or MRI positive lesions to biopsy histopathology, cancer grade group, PSA and other clinical parameters | one study visit (up to 3.5 hours)
  Qualitative and quantitative PET and MRI parameters for PET and/or MRI positive lesions will be correlated with biopsy histopathology, cancer grade group, PSA and other clinical parameters.
Sub-study 4: Change in Gleason Score | one study visit (up to 3.5 hours), post-prostatectomy (standard of care)
  PET and MRI directed biopsy histopathology prostate Gleason score range will be compared, and evaluated for Gleason score upgrading in any patients who undergo prostatectomy with available prostatectomy histopathology as the reference standard. Gleason scores range from 6-10 with higher numbers indicating higher grade cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Y Cho, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/